CLINICAL TRIAL: NCT04540809
Title: Effect of Psoriatic Arthritis on the Strength, Proprioception, Skill, Coordination, and Functional Condition of the Hand
Brief Title: The Effect of Psoriatic Arthritis on the Functions of the Hand
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burcu Talu, Associate Professor, Inonu University
Other Study IDs: 2019 / 7-21
Record Dates: First submitted 2020-08-28; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Psoriatic Arthropathy Hand; Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Pathogenesis; Disease activity; Hand
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Proprioception

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psoriatic arthritis group (PsAG): The evaluation was made using dynamometer, goniometer, mobile application, and Purdue pegboard test.
  Interventions: Other: Assessment of strength, proprioception, skill and coordination of the hand

INTERVENTIONS:
Other: Assessment of strength, proprioception, skill and coordination of the hand — Disease Activity Score 28 was used to determine the disease activity of patients with PsA. Grip strength was measured with the help of Baseline Digital Hand Dynamometer®. Pinch strength was measured with Baseline Hydraulic Pinch Gauge®. Wrist proprioception was assessed by measuring the joint position sensation using a goniometer by actively repeating the target angle predetermined by the researcher (30 ° for flexion and extension, 15 ° for ulnar deviation, 10 ° for radial deviation. Finger skills were assessed using a mobile application called Ball Tap©. The application included the fastest contact of the participants to the balls coming from different parts of the screen for 30 seconds. Two hand coordination and skills were evaluated using the Purdue Pegboard test. The Michigan Hand Outcomes Questionnaire was used for functional evaluation of the hand, and the Health Assessment Questionnaire was used to assess the general functional condition and health-related quality of life.

SUMMARY:
This study was planned to evaluate the effect of psoriatic arthritis on the strength, proprioception, skill, coordination, and functional condition of the hand and to determine the correlate disease activity with these parameters.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is a chronic, progressive, inflammatory arthritis that occurs as a condition associated with patients with psoriasis and may result in permanent joint damage and an increased risk of mortality. Synovial membrane inflammation characterized by increased vascularization and immune cell infiltration is an important feature of psoriatic arthritis. This inflamed synovial microenvironment leads to the formation of synovial pannus, entheseal inflammation, and joint damage. Although PsA is generally thought of as a benign arthropathy, structural damage has been shown with the progression of the disease, along with joint inflammation.As a result of the researches, it has been stated that tissue biomechanical stress and microtraumas that lead to the activation of abnormal natural immune responses in psoriatic arthritis can trigger joint inflammation. In parallel, inflammation is expected to be more common in peripheral joints, which are known to be more exposed to microtrauma. Studies have reported that hand joint involvement is frequently seen in patients with PsA and is an important cause of loss of function and that erosions in hand joints are associated with statistically significant loss of hand strength. Theoretically, either the mechanical effect of the fluid in the acute joint effusion or the components of the inflammatory fluid and the changing capsular compliance after chronic effusion and has been reported that problems may occur in proprioception due to causes such as pain, trauma, and fatigue. However, pain, decreased joint ROM and grip strength, muscle weakness, and hand deformities can affect hand fine hand skills and function. The hypothesis of this study is that supporting the clinical condition of the participants with parameters related to general hand function will be effective in predicting disease progression and disability. Accordingly, the aim of the researchers is to evaluate the effect of PsA on the grip and pinch strength of the hand, proprioception, skill, coordination and functional status, and to determine the relationship of disease activity with these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-65

Exclusion Criteria:

* Neurological diseases that caused sequelae at hand, upper extremity surgeries, neuropathies, traumas, and history of nerve damage
* Psychiatric disorders,
* Reluctance to continue evaluation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals and healthy controls diagnosed with PsA according to the classification criteria for PsA (Classification Criteria for Psoriatic Arthritis, CASPAR).
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Handgrip strength | 3 months
  Handgrip was measured with the Baseline Digital Hand Dynamometer 135 KG®. The results were recorded as Kg.
Pinch strength | 3 months
  Pinch strength was measured with the Baseline Hydraulic Compaction Meter 45 KG®. The results were recorded as Kg.
Wrist proprioception | 3 months
  Wrist proprioception was assessed by measuring joint position sense with a goniometer. Error average of 3 repetitions in each movement axis was recorded. Low scores indicate a better functional status.
Finger skills | 3 months
  Finger skills were recorded as points at the end of 30 seconds with the mobile application. Higher scores indicate better functional status.
Both hand skill and coordination | 3 months
  Both hand skill and coordination were evaluated using the Purdue Pegboard test. It consists of 4 parts. These; right and left hand, both hands, and assembly. Higher scores indicate better function.

SECONDARY OUTCOMES:
Disease activity | 3 months
  DAS28 is a measurement method that determines the disease activity by using the number of painful and swollen joints, ESR (erythrocyte sedimentation rate) or C-reactive protein values in the first hour, and a 100 mm visual analog scale for general evaluation. ESR was used in this study. Higher scores indicate higher disease activity.
Michigan Hand Outcomes Questionnaire | 3 months
  The MHQ is a self-report measure that assesses the function of hand (s) and / or wrist (s). The MHQ contains six distinct scales including overall hand function, activities of daily living, pain, work performance, aesthetics and subject satisfaction with hand function. Each question is scored on a scale of 1-5. High score in total scores indicates high satisfaction.
Health Assessment Questionnaire | 3 months
  It is a questionnaire consisting of 8 subtitles evaluating daily life activities. Each question ranges from zero (no functional impairment) to three (task disabling). Points between 0-60 are received.Lower scores indicate better conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu TALU, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No